CLINICAL TRIAL: NCT02095275
Title: Exploring the Relationship Among Brain Natriuretic Peptide, Fluid Status and Acute Kidney Injury in Critically Ill Patients
Brief Title: Exploring the Relationship Among BNP, Fluid Status and Acute Kidney Injury in Critically Ill Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201111012RIB
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Acute Kidney Injury (Nontraumatic)
Keywords: BNP, acute kidney injury, fluid status
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum BNP
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute kidney injury: ICU patients with Acute kidney injury

SUMMARY:
B-type natriuretic peptide (BNP) is rapidly released by the ventricles of the heart in response to myocardial stretch. This cardiac neurohormone is mostly elevated in patients with fluid overload or myocardium dysfunction. BNP is a very useful and important marker. It can predict mortality and cardiac events in patients in the ICU setting. In stable hemodialysis patients with normal LV function on echocardiography, high BNP levels are likely the result of blood volume expansion and require reduction in postdialysis dry weight.

In the past, there were many methods to evaluate fluid status. Some are not reliable such as central venous pressure or physical examination. Some are invasive and expensive such as Swan Ganz、PiCCO catheter or bioimpedance device. Nevertheless, About the relationship between BNP and fluid status, a study found a significant relation between bioimpedance-derived body composition (BC) (fluid distribution) parameters and BNP concentrations. This relationship was independent of the cardiac history of the patient and suggests that the natriuretic peptide levels are to some degree modifiable by changing a patient's fluid distribution.

In this study, the investigators want to observe that if the level of BNP can predict the occurrence of acute kidney injury and the need of renal replacement therapy. Besides, the investigators also want to see if BNP can be a useful and convenient marker to guide adjustment of optimal fluid status and then to improve outcome.

DETAILED DESCRIPTION:
B-type natriuretic peptide (BNP) is rapidly released by the ventricles of the heart in response to myocardial stretch. This cardiac neurohormone is mostly elevated in patients with fluid overload or myocardium dysfunction. BNP is a very useful and important marker. It can predict mortality and cardiac events in patients in the ICU setting. In stable hemodialysis patients with normal LV function on echocardiography, high BNP levels are likely the result of blood volume expansion and require reduction in postdialysis dry weight.

On the other hand, ample recent data have highlighted the role of ﬂuid accumulation on mortality and non-recovery of kidney function in critically ill patients with acute kidney injury (AKI). In the past, there were many methods to evaluate fluid status. Some are not reliable such as central venous pressure or physical examination. Some are invasive and expensive such as Swan Ganz、PiCCO catheter or bioimpedance device. Nevertheless, About the relationship between BNP and fluid status, a study found a significant relation between bioimpedance-derived body composition (BC) (fluid distribution) parameters and BNP concentrations. This relationship was independent of the cardiac history of the patient and suggests that the natriuretic peptide levels are to some degree modifiable by changing a patient's fluid distribution.

In this study, we want to observe that if the level of BNP can predict the occurrence of acute kidney injury and the need of renal replacement therapy. Besides, we also want to see if BNP can be a useful and convenient marker to guide adjustment of optimal fluid status and then to improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 y/o in ICU

Exclusion Criteria:

* Acute coronary syndrome
* Congestive heart failure history
* Clinical pulmonary hypertension with various cause (iPAH, congenital heart disease, CTEPH, COPD with cor pulmonate,…)
* Patients with acute pulmonary embolism
* Chronic atrial fibrillation,
* Respiratory failure with high PEEP (>10 CmH2)
* Terminal cancer patients
* Patients with Bosmina therapy
* Patients received CPR (IHCA or OHCA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in intensive care unit(older than 18 y/o)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in serum creatinine level at 3 months | 3 months

SECONDARY OUTCOMES:
Mortality | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Hsiang Chou, bachelor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan